CLINICAL TRIAL: NCT03760536
Title: Get REAL and HEEL Research Program
Status: Completed | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: LCCC 1630
Record Dates: First submitted 2018-10-22; First posted 2018-11-30 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Blood draw for p16 analysis and immune/inflammatory parameters
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 16-week Exercise Program: Interested patients will attend a group meeting where they will be screened and consented to the study. During weeks 1 and 2 patients will complete pre-intervention baseline assessments and blood draws followed by a 16-week supervised exercise program at Get REEL and HEAL facility. Study participants will complete progressive aerobic and resistance exercise training. Post-intervention weeks 1 and 2 participants will complete assessments, questionnaires and blood draws. Participants will be followed up at 6 and 12 months post intervention with physical assessments, questionnaires and blood draws. Annual follow-up will occur at year 2,3,4 and 5 post intervention with questionnaires only.
  Interventions: Behavioral: 16-week Exercise Rehabilitation Program for Breast Cancer Survivors

INTERVENTIONS:
Behavioral: 16-week Exercise Rehabilitation Program for Breast Cancer Survivors — Interested patients will attend a group meeting where they will be screened and consented to the study. During weeks 1 and 2 patients will complete pre-intervention baseline assessments and blood draws followed by a 16-week supervised exercise program at Get REEL and HEAL facility. Study participants will complete progressive aerobic and resistance exercise training. Post-intervention weeks 1 and 2 participants will complete assessments, questionnaires and blood draws. Participants will be followed up at 6 and 12 months post intervention with physical assessments, questionnaires and blood draws. Annual follow-up will occur at year 2,3,4 and 5 post intervention with questionnaires only.

SUMMARY:
The UNC Get REAL & HEEL (GR&H) program has provided after treatment support for women with a breast cancer diagnosis since 2006. The 16-week program includes an individualized training program and the opportunity to continue working out in the GR&H facilities at the conclusion of the 16-week program. The purpose of this protocol is to implement a research agenda at GR&H that will examine the efficacy of the program. The primary aim of this study is a pre-post test of the impact of the GR&H program (standardized combination of aerobic and resistance training) on VO2peak1,2. The secondary aims of this study are to evaluate quality of life as well as cardiorespiratory function (vascular health), physical function (muscular strength, body composition), cognition, balance, and patient-reported outcomes (fatigue, depression, anxiety, quality of life). Exploratory aims are focused on evaluating the impact of exercise on biomarkers: (1) aging - p16INK4a, (2) immune cell function - total leukocyte count, T and natural killer cells, monocytes, and neutrophils count and activity, and (3) circulating pro- and anti-inflammatory cytokines.

DETAILED DESCRIPTION:
Objectives:

Primary:

Evaluate the impact of the Get REAL and HEEL research program (standardized combination of aerobic and resistance training) on change in V02peak from pre to post 16-week intervention.

Secondary:

Evaluate the impact of the GR&H program (standardized combination of aerobic and resistance training) on change in cardiorespiratory function, immunology, physical function parameters, cognition, balance, and patient-reported outcomes from pre to post 16-week intervention.

Evaluate changes in all measures annually over the 5 year follow-up period.

Report on enrollment, recruitment, and attrition.

Exploratory Objectives

The investigator's exploratory aims are focused on evaluating the impact of exercise on biomarkers: (1) aging - p16INK4a, (2) total leukocyte, lymphocyte (T cells and natural killer cells), monocyte and neutrophil counts and T cell proliferation assays, natural killer cytotoxicity assays, and cytokine production from stimulated neutrophils and monocytes, and (3) circulating pro- and anti-inflammatory cytokines.

OUTLINE:

Participants will complete pre-intervention assessments, questionnaires and blood draw at week 1 and 2 pre-intervention, followed by a 16-week aerobic and resistance training exercise program (intervention). Participants will complete assessments, questionnaires and blood draws at week 1 and 2 following the intervention and then again at 6 months and 12 months following intervention. Questionnaires only will be administered at year 2, 3,4 and 5 following intervention.

ELIGIBILITY:
Inclusion Criteria:

Patients will be eligible for this protocol if they have

* histologically confirmed early stage (non-metastatic) breast cancer
* and have recently (within 1 year) completed their initial treatment (they may continue to be on endocrine treatment).

No exclusions will be made based on ethnicity or race, although patients must be able to read and speak English.

Participants must provide IRB-approved signed written informed consent. The consent includes access to their medical records, including demographic and billing information, diagnoses, treatments, and laboratory results. Participants may also be asked to provide permission to contact their non-UNC doctors for additional medical record information, and may also require a medical release from various treating physicians.

Interested persons must agree to adhere to the 16-week GR&H protocol and complete all blood draws, assessments and questionnaires to the best of their ability. The informed consent will also include annual follow-up assessments and questionnaires for up to 5 years after they have completed the 16-week program.

Patients who are approached about participating in LCCC1630 and decline to do so are able to join GR&H as a supportive care program.

Exclusion Criteria:

Interested persons will be excluded from study participation if

* they do not have evidence of a cancer diagnosis or completion of surgery, radiation and/or chemotherapy treatment,
* or if they have previously completed the GR&H exercise program. Entirely at the discretion of GR&H investigators, physical function and other assessments conducted at baseline may also determine that a patient is not medically suitable for the GR&H protocol. Consented patients who are determined to be medically not suited for the GR&H protocol (unevaluable) will remain in the study for analyses comparing those who are evaluable with those who are not.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential study participants with confirmed early-stage breast cancer will be screened through a review of daily clinic schedules for patients seen at the North Carolina Cancer Hospital. Patients must have recently completed their initial treatment (be within one year of completion).
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2019-03-09 (Actual); Study Completion 2020-02-12 (Actual)

PRIMARY OUTCOMES:
Cardiopulmonary exercise test with NIRS and PWA (vascular function) | Pre-intervention (weeks 1-2), Post-intervention (weeks 17 or 18), 6 months post-intervention, 12-months post intervention
  The Cardiopulmonary Exercise Test (CPET) with NIRS and PWA will be used to measure peak oxygen content (VO2peak), tissue oxygen saturation and pulse wave analysis during this symptom-limited exercise test.

SECONDARY OUTCOMES:
Anthropometrics-Height | Pre-intervention (weeks 1-2), post-intervention (weeks 17 or 18), 6 months post intervention, 12 months post-intervention
  Measure Height
Anthropometrics-Weight | Pre-intervention (weeks 1-2), post-intervention (weeks 17 or 18), 6 months post intervention, 12 months post-intervention
  Weight
Anthropometrics-BMI | Pre-intervention (weeks 1-2), post-intervention (weeks 17 or 18), 6 months post intervention, 12 months post-intervention
  Measure BMI
Anthropometrics-Blood Pressure | Pre-intervention (weeks 1-2), post-intervention (weeks 17 or 18), 6 months post intervention, 12 months post-intervention
  Measure blood pressure -- both systolic and diastolic
Anthropometrics-Resting Heart Rate | Pre-intervention (weeks 1-2), post-intervention (weeks 17 or 18), 6 months post intervention, 12 months post-intervention
  Measure Resting Heart Rate
Body Composition | Pre-intervention (weeks 1-2), post-intervention (weeks 17 or 18), 6 months post-intervention, 12 months post-intervention
  DEXA -- Body Composition will be perfomed using a Hologic (Discovery W) Dual X-ray Absorptiometry (DEXA) located in the EORL. Total body weight-mass (BW) and compositional aspects of lean body mass (LBM), fat tissue mass (FM), and percentage body fat (% BF) will be examined using standard DEXA screening procedures. The BW will be measured using a high grade analytical balance-scale (accuracy ± 10 grams).
Measure of muscle composition -- proportion of body fat to lean muscle mass | Pre-intervention (weeks 1-2), post-intervention (weeks 17 or 18), 6-months post-intervention, 12-months post-intervention
  Ultrasound -- LogicView™ software (General Electric Company, Milwaukee, WI, USA) will be used to generate real-time panoramic cross-sectional images of the VL. Three panoramic scans at a gain of 50dB and a depth of 5.0 cm. All image analyses will be completed using Image-J software (version 1.46r, National Institutes of Health, USA) with each image area individually scaled from pixels to centimeters via the straight-line function. The polygon function will be used to determine the CSA of the VL by selecting a region including mostly muscle and minimal surrounding fascia. Greater EI values represent greater fibrous (non-muscular) composition.
Vascular Function | Pre-intervention (weeks 1-2), post-intervention (weeks 17 or 18), 6-months post-intervention, 12-months post-intervention
  XCEL Sphygmacor+USCOM
Resting ECG | Pre-intervention (weeks 1-2), post-intervention (weeks 17 or 18), 6-months post-intervention, 12-months post-intervention
  Resting electrocardiogram -- Individual wave/complex/intervals components and overall ECG tracings will be assessed using a 12-lead ECG. The study Cardiologist will review each report individually at baseline prior to the Cardiopulmonary Exercise Test for evidence of overt cardiac dysfunction and will deem the potential study participant appropriate/not appropriate for exercise testing.
Functional Tests | Pre-intervention (weeks 1-2), post-intervention (weeks 17 or 18), 6-months post-intervention, 12-months post-intervention
  6-minute walk
Functional Tests | Pre-intervention (weeks 1-2), post-intervention (weeks 17 or 18), 6-months post-intervention, 12-months post-intervention
  Timed Up and Go
Cognitive Testing | Pre-intervention (weeks 1-2), post-intervention (weeks 17 or 18), 6-months post-intervention, 12-months post-intervention
  Administer DKEFS
Cognitive Testing | Pre-intervention (weeks 1-2), post-intervention (weeks 17 or 18), 6-months post-intervention, 12-months post-intervention
  Administer Digit Span
Cognitive Testing | Pre-intervention (weeks 1-2), post-intervention (weeks 17 or 18), 6-months post-intervention, 12-months post-intervention
  Administer Sequencing
Cognitive Testing | Pre-intervention (weeks 1-2), post-intervention (weeks 17 or 18), 6-months post-intervention, 12-months post-intervention
  Administer HVLT-R
Cognitive Testing | Pre-intervention (weeks 1-2), post-intervention (weeks 17 or 18), 6-months post-intervention, 12-months post-intervention
  Administer TMT
Cognitive Testing | Pre-intervention (weeks 1-2), post-intervention (weeks 17 or 18), 6-months post-intervention, 12-months post-intervention
  Administer NeuroCom balance test
Muscle Strength and Power | Pre-intervention (weeks 1-2), post-intervention (weeks 17 or 18), 6-months post-intervention, 12-months post-intervention
  Isokinetic, isometric handgrip tests
Blood Draw | Pre-intervention (weeks 1-2), post-intervention (weeks 17 or 18), 6-months post-intervention, 12-months post-intervention
  30 mL Blood draw for non-subset group
Satisfaction with GR&H Questionnaire | Pre-intervention (weeks 1-2), post-intervention (weeks 17 or 18), 6-months post-intervention, 12-months post-intervention
  Administer Satisfaction with GR&H Questionnaire
Acute exercise bout with blood draw for immune/inflammatory parameters (subset group only) | Pre-intervention (weeks 1-2), post-intervention (weeks 17 or 18), 6-months post-intervention, 12-months post-intervention
  Cannulated, 3 blood draws over course of 45 minute visit. 50 mL total collected pre-intervention and post intervention; 30 mL total collected at 6 months and 12 months post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Claudio L Battaglini, PhD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center; Kirsten Nyrop, Study Director — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- North Carolina Cancer Hospital, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Wagoner CW, Lee JT, Hanson ED, Kerr ZY, Nyrop KA, Muss HB, Battaglini CL. Baseline fatigue in early breast cancer survivors: understanding its prevalence in community-based exercise. Support Care Cancer. 2022 May;30(5):4407-4416. doi: 10.1007/s00520-021-06776-8. Epub 2022 Jan 31. PMID 35098347
- [Derived] Bartlett DB, Hanson ED, Lee JT, Wagoner CW, Harrell EP, Sullivan SA, Bates LC, Alzer MS, Amatuli DJ, Deal AM, Jensen BC, MacDonald G, Deal MA, Muss HB, Nyrop KA, Battaglini CL. The Effects of 16 Weeks of Exercise Training on Neutrophil Functions in Breast Cancer Survivors. Front Immunol. 2021 Oct 27;12:733101. doi: 10.3389/fimmu.2021.733101. eCollection 2021. PMID 34777343
- [Derived] Hanson ED, Bates LC, Harrell EP, Bartlett DB, Lee JT, Wagoner CW, Alzer MS, Amatuli DJ, Jensen BC, Deal AM, Muss HB, Nyrop KA, Battaglini CL. Exercise training partially rescues impaired mucosal associated invariant t-cell mobilization in breast cancer survivors compared to healthy older women. Exp Gerontol. 2021 Sep;152:111454. doi: 10.1016/j.exger.2021.111454. Epub 2021 Jun 16. PMID 34146655